CLINICAL TRIAL: NCT04582136
Title: Efficacy and Safety of Sirolimus in Patients With Active Systemic Lupus Erythematosus Despite Standard of Care: a Multi-center, Double Blinded, Randomized, Placebo-controlled, Phase 3 Trial
Brief Title: Efficacy and Safety of Sirolimus in Active Systemic Lupus Erythematosus
Acronym: SIRIUS
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Chinese SLE Treatment And Research Group (Other)
Collaborators: Beijing Municipal Science & Technology Commission (Other); North China Pharmaceutical Group Corporation (Industry)
Responsible Party: Principal Investigator, Xiaofeng Zeng, Director of Rheumatology and Immunology Department Chinese Academy of Medical Sciences &Peking Union Medical College Hospital, Chinese SLE Treatment And Research Group
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CSTAR_RCT_SLE_001
Record Dates: First submitted 2020-10-03; First posted 2020-10-09 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Systemic Lupus Erythematosus
Keywords: mTOR; systemic lupus erythematosus; SLE; lupus erythematosus; sirolimus; rapamycin
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — Sirolimus

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sirolimus plus SOC (Experimental): Sirolimus plus standard therapy (SOC) for SLE; Generic name: sirolimus (0.5mg capsule); Dosage: 1.5mg/day; Administration route: Oral
  Interventions: Drug: Sirolimus
- Placebo plus SOC (Placebo Comparator): Placebo plus standard therapy (SOC) for SLE; Drug: Placebo comparator plus SOC; Administration route: Oral
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Sirolimus — In the double-blinded phase, sirolimus 1.5mg/day plus SOC is administered throughout 24 weeks; in the open-label extension period, patients who opt to participate continue on sirolimus 1.5mg/day plus SOC for an additional 24 weeks.
  Other Names: rapamycin
  Arms: Sirolimus plus SOC
Drug: Placebo — In the double-blinded phase, placebo plus SOC is administered throughout 24 weeks; in the open-label extension period, patients who opt to participate are switched to receive sirolimus 1.5mg/day plus SOC for an additional 24 weeks.
  Arms: Placebo plus SOC

SUMMARY:
This is a multi-center, double-blinded, randomized, placebo-controlled, phase 3 study to evaluate the efficacy and safety of sirolimus administered in addition to standard therapy, in patients with active SLE disease.

DETAILED DESCRIPTION:
This study is a multi-center, double-blinded, randomized, placebo-controlled, phase 3 clinical trial to assess the efficacy and safety of sirolimus in patients with active systemic lupus erythematosus despite receiving standard background therapy.

Six large rheumatological referring centers across from China will participate in the study.

The study is divided into two phases. The first phase is a 24-week randomized, double-blinded, placebo-controlled trial, from which the primary end point will be generated, and the second phase is a 24-week open-labeled extension trial.

The study enrolls SLE patients between 18~65 years old who have SLEDAI-2K score ≥4 (not including scores for anti-dsDNA antibody and hypocomplementemia), despite conventional treatment (e.g., immunosuppressants, antimalarial drugs, glucocorticoids, NSAIDs, anti-hypertensive drugs, and/or topical medications). In addition, subjects must be serologically active (positive anti-dsDNA antibody and/or hypocomplementemia).

Subjects will be randomly assigned by 1:1 ratio to receive sirolimus (1.5mg/day) or placebo for the first 24-week phase. In the second 24-week open-labeled phase, sirolimus patients receive the same dose of sirolimus, and placebo group are switched to receive sirolimus at 1.5mg/day

ELIGIBILITY:
Inclusion Criteria:

* Age between 18~65 years;
* Fulfilling the 2012 SLICC criteria for SLE; time from SLE diagnosis ≥ 3 months;
* Active disease as defined by a SLEDAI-2K score of ≥4 (not including scores for anti-dsDNA antibody and hypocomplementemia) at screening;
* Serologically active defining as positive anti-dsDNA antibody (>10IU/ml) or hypocomplementemia (C3<0.90g/L)
* Before the first dose of sirolimus, a stable regimen of oral corticoids (0-20 mg/day, prednisone or equivalent) ≥4 weeks; doses of antimalarials, or immunosuppressive agents (mycophenolate mofetil [MMF]/mycophenolic acid [MPA] ≤1.5g/day, or MTX ≤15mg/week) are required to be stable for at least 12 weeks prior to first dose). In addition, angiotensin-converting enzyme inhibitors or angiotensin receptor blockers, NSAIDs or other analgesics should be stable for at least 2 weeks.

Exclusion Criteria:

* Concomitant connective tissue disease or inflammatory disease that might confound efficacy assessments, e.g., systemic sclerosis, rheumatoid arthritis, dermatomyositis/polymyositis, etc;
* Neuropsychiatric SLE;
* Severe active lupus nephritis (urinary protein ≥3.5g/24h or urine protein/creatine ration> 3500mg/g or eGFR < 60ml/1.73m2/min);
* Pregnant or breast-feeding women;
* Previous treatment with sirolimus or allergic to sirolimus;
* Intravenous CTX within 6 months of enrollment;
* Intravenous immunoglobulin or prednisone dose >100mg/day within 3 months;
* Calcineurin inhibitors (e.g., tacrolimus or cyclosporin A) within 1 month;
* Traditional Chinese Herb (such as Tripterygium wilfordii Hook F) within 1 month;
* Concurrent active or uncontrolled infection (such as tuberculosis and hepatitis) requiring antibiotics or antivirus;
* WBC count <3×10^9/L;
* Abnormal biochemical indices including: alanine transaminase (ALT) or aspartate aminotransferase (AST) >1.5 times upper limit of laboratory reference range; total bilirubin or blood lipid (including total cholesterol, triglycerides, and low-density lipoprotein) >2 times upper limit of laboratory reference range;
* Any condition that may require multiple courses of systemic corticosteroids (e.g., uncontrolled asthma, COPD);
* Major surgery within the past month;
* Suffering from malignant tumors or a history of malignant tumors within 5 years before screening, or a history of lymphoproliferative diseases: Patients with previously treated cutaneous squamous cell carcinoma and basal cell carcinoma without evidence of recurrence are allowed to enroll; and Patients with cervical cancer in situ who have documented formal surgical cure are allowed to enroll;
* Previous stem cell transplantation (including hematopoietic stem cell transplantation and mesenchymal stem cell transplantation);
* Have a history of splenectomy;
* Subjects has certain conditions that may lead to dropping out of the study in advance or that may bring risk to subjects themselves if they participate in the study. This is judged by experienced clinicians.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 146 (Estimated)
Dates: Start 2021-03-04 (Actual); Primary Completion 2025-04-21 (Actual); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
The Proportion of Patients Who Achieve an SLE Responder Index-4 (SRI-4) Composite Response at Week 24 | 24 weeks
  SLE responder index-4 (SRI-4), is a composite outcome includes all of the following outcomes: a reduction of SLEDAI-2K ≥ 4 points, no new BILAG A organ domain scores and no more than 1 new BILAG B organ domain scores, and no worsening of PGA (increase < 0.3).

SECONDARY OUTCOMES:
Change From Baseline in Complement Level at Week 24 | 24 weeks
  Serum complement refers to C3 and C4, which are both detected in the central lab.
Change From Baseline in Titers of Anti-dsDNA Antibody at Week 24 | 24 weeks
  Anti-dsDNA antibody is detected in the central lab using chemiluminescence.
Change From Baseline in Systemic Lupus Erythematosus Disease Activity Index 2000 (SLEDAI-2K) Score at Week 24 | 24 weeks
  The SLEDAI-2K is an established, validated SLE activity index. It is based on the presence of 24 features in 9 organ systems and measures disease activity in SLE patients in the previous 30 days. It is weighted according to the feature. Features are scored by the assessing physician if present within the last 30 days with more severe features having higher scores, and then simply added to determine the total SLEDAI 2K score, which ranges from 0 to 105, with higher scores representing increased disease activity.
Change From Baseline in Physician's Global Assessment of Disease Activity (PGA) Score at Week 24 | 24 weeks
  PGA is recorded on a visual analogue scale (VAS; 0.0 to 10.0 centimeter [cm]). The scale for the physician's assessment ranges for 'no lupus activity' (0.0) to 'extremely active lupus' (10.0).
Number of Participants With BILAG-based Combined Lupus Assessment (BICLA) Response at Week 24 | 24 weeks
  BICLA response defined as participants meeting following criteria: 1. BILAG improvement (all BILAG A scores at baseline improved to either B, C or D and all BILAG B scores at baseline improved to C or D and no worsening in disease activity defined as no new BILAG A scores and <= 1 new BILAG B score) and 2. no worsening of total SLEDAI-2K from baseline 3. < 1 cm increase in PGA and 4. no treatment failure criteria met. BILAG: assesses disease extent, severity (range: A [severe] to E [no disease]). SLEDAI-2K: assesses improvement in disease activity (range: 0 to 105; higher score = higher severity). PGA: assesses worsening in participant's general health status (0.0= 'no lupus activity' to 10.0 = 'extremely active lupus').

OTHER OUTCOMES:
Change From Baseline in SLE Disease Activity Score (SLE-DAS) at Week 24 | 24 weeks
  SLE-DAS is a newly developed tools to assess SLE disease activity. It is a multinomial that includes 17 clinical or laboratory indices: arthritis, swollen joint count, mucocutaneous vasculitis, localized cutaneous rash, generalized cutaneous rash, alopecia, mucosal ulcers, hypocomplementaemia, increased anti-dsDNA antibody, proteinuria, thrombocytopenia, leucopenia, neuropsychiatric involvement, systemic vasculitis, cardiac/pulmonary involvement, myositis, serositis, and haemolytic anaemia.The SLE-DAS is a continuous disease activity score with higher values signifying greater disease activity.
Percentage of Patients With Clinical Remission at week 24 | 24 weeks
  Clinical remission is defined as clinical SLEDAI-2K (cSLEDAI-2K, excluding items from hypocomplementemia or positive anti-dsDNA antibody) = 0 AND that allowable dose of glucocorticoids is ≤ 5 mg/day prednisone (or equivalent)
Percentage of Patients With Lupus Low Disease Activity State (LLDAS) at week 24 | 24 weeks
  LLDAS is defined as: (1) SLE Disease Activity Index (SLEDAI)-2K ≤4, with no activity in major organ systems (renal, central nervous system (CNS), cardiopulmonary, vasculitis, fever) and no haemolytic anaemia or gastrointestinal activity; (2) no new lupus disease activity compared with the previous assessment; (3) a Safety of Estrogens in Lupus Erythematosus National Assessment (SELENA)-SLEDAI physician global assessment (scale 0-3) ≤1; (4) a current prednisolone (or equivalent) dose ≤7.5 mg daily; and (5) well tolerated standard maintenance doses of immunosuppressive drugs and approved biological agents.
Percentage of Patients With Hypocomplementemia returned to normal at week 24 | 24 weeks
  Percentage of patients whose hypocomplementemia are returned to normal (C3>0.90g/L AND C4>0.10g/L)
Percentage of Patients With Anti-dsDNA Antibody decreased to negative at week 24 | 24 weeks
  Percentage of Patients With Anti-dsDNA Antibody decreased to <10 IU/ml.
Change From Baseline in Urine Protein/Creatine Ratio (PCR) Among Patients With Baseline PCR >500mg/g at Week 24 | 24 weeks
  PCR is detected in the central lab
The Time to First BILAG Flare | 24 weeks
  First BILAG flare is defined as at least one new BILAG A score or at least two new BILAG B scores
Proportions of Patients With an SRI-5 and SRI-6 Response at Week 24 | 24 weeks
  The definitions of SRI-5 and SRI-6 is similar with SRI-4 except for a reduction of SLEDAI-2K ≥ 5 points or ≥ 6 points respectively
Proportion of Patients With No Worsening in BILAG at Week 24 | 24 weeks
  No worsening in BILAG is defined as no new BILAG A score and no more than one new BILAG B score
Proportions of Patients With No Worsening in PGA at Week 24 | 24 weeks
  No increase in PGA scores
Change From Baseline in 36-Item Short Form Survey (SF-36) | 24 weeks
  As a concise health questionnaire, SF-36 comprehensively summarizes the quality of life of the subjects from eight aspects: physiological function, physiological function, physical pain, general health status, energy, social function, emotional function and mental health. SF-36 scores range from 0 (maximum disability) to 100 (no disability).
Change From Baseline in Lupus Patient-Reported Outcome tool (LupusPRO) | 24 weeks
  LupusPRO is a valid and reliable patient-reported health outcome targeting towards measuring health (HRQOL) and non-health related quality of life (Non HRQOL) among patients with systemic lupus erythematosus (SLE). It assess the quality of life from 14 aspects: lupus symptoms, cognition, lupus medications, procreation, physical health, sleep, vitality, pain, emotional health, body image, desires-goals, social-support, coping, satisfaction with care. The score range of LupusPRO is from 0 to 100 points, where higher scores represent better quality of life, while lower scores indicate poorer quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaofeng Zeng, MD, Principal Investigator — Chinese SLE Treatment and Registration Group
Locations (6):
- China (6):
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - Shenzhen People's Hospital, Shenzhen, Guangdong
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - The Second Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - The First Hospital of China Medical University, Shenyang, Liaoning
  - First Affiliated Hospital of Kunming Medical University, Kunming, Yunnan

IPD SHARING:
Plan to Share IPD: Yes
all IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: IPD will be available when the study result is published.